CLINICAL TRIAL: NCT03382912
Title: A Randomized Phase 2 Trial of AM0010 in Combination With Nivolumab vs. Nivolumab Alone as Second-Line Therapy in Subjects With Stage IV / Metastatic Wild Type Non-Small Cell Lung Cancer and Low Tumor Expression of PD-L1
Brief Title: Study of Pegilodecakin (LY3500518) With Nivolumab Compared to Nivolumab Alone Second-line Tx in Participants With Metastatic Non-Small Cell Lung Cancer
Acronym: Cypress 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The CYPRESS-2 trial was closed early after the planned final analysis because the risk benefit ratio is unfavorable.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17161; J1L-AM-JZGD (Other: Eli Lilly and Company); AM0010-202 (Other: ARMO BioSciences)
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pegilodecakin; AM0010; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegilodecakin+Nivolumab (Experimental): Participants received Pegilodecakin subcutaneously at 0.8 milligrams (mg) (≤80 kilograms (kg) body weight) or 1.6 mg (>80 kg body weight) once daily (QD) in the abdomen, thigh or back of upper arm.
  Nivolumab administered on day 1 of each 14 or 28 day cycle over approximately 30 minutes intravenous (IV) infusion at 240 mg every 2 weeks (Q2W), or 480 mg every 4 weeks (Q4W).
  Interventions: Biological: Pegilodecakin; Drug: Nivolumab
- Nivolumab (Active Comparator): Participants received Nivolumab on day 1 of each 14- or 28- day cycle over approximately 30 minutes intravenous (IV) infusion at 240 mg every two weeks (Q2W), or 480 mg every 4 weeks (Q4W).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Biological: Pegilodecakin — Pegilodecakin plus Nivolumab
  Other Names: LY3500518; AM0010
  Arms: Pegilodecakin+Nivolumab
Drug: Nivolumab — Nivolumab Alone

SUMMARY:
To compare the efficacy of pegilodecakin in combination with nivolumab versus nivolumab alone in participants with metastatic non-small cell lung cancer as measured by objective response rate.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, Phase 2 study designed to compare the efficacy and safety of pegilodecakin in combination with nivolumab versus nivolumab alone in participants with stage IV / metastatic wild type non-small cell lung cancer and tumors with low tumor expression of PD-L1 (0-49%).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed Wild Type NSCLC that is stage IV / metastatic or recurrent
2. Participants must have received at least one prior systemic therapy that was not an anti-PD-1, anti-PD-L1 and/or anti-CTLA-4 treatment for the advanced stage of the disease
3. Participants with tumor tissue low expression of PD-L1 as defined by Tumor Proportion Score (TPS) 0% - 49%
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Participants with measurable disease by spiral computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumor (RECIST) v.1.1 criteria
6. Participants that have completed prior radiotherapy or radiosurgery at least 2 weeks prior to randomization

Exclusion Criteria:

1. Participants with active central nervous system (CNS) metastases or carcinomatous meningitis
2. Participants with any serious or uncontrolled medical disorder or active infection with the hepatitis virus or the human immunodeficiency virus (HIV)
3. Participants with Grade 1 (NCI-CTCAE v.4.03) toxicities attributed to prior anti-cancer therapy (other than alopecia and fatigue) prior to randomization
4. Participants that have received nivolumab
5. Participants that have received therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents
6. Participants with a history of severe hypersensitivity reactions to monoclonal antibodies
7. Participants that have received therapy with anti-PD-1, anti-PD-L1, anti-PD-L-2, anti-CD-137, and/or anti CTLA-4 antibodies
8. Participants receiving any investigational agent within 28 days of first administration of trial treatment
9. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (35):
  - Arizona Oncology Associates, P.C., Tempe, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Glendale Adventist Medical Center, Los Angeles, California
  - Redwood Regional Oncology Center, Santa Rosa, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Center, Lone Tree, Colorado
  - John B. Amos Cancer Center, Columbus, Georgia
  - Covenant Clinic, Waterloo, Iowa
  - Baptist Health Medical Group, Lexington, Kentucky
  - MedStar Health Research Institute, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Sparrow Health System, Lansing, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Valley Hospital - Luckow Pavilion, Westwood, New Jersey
  - Broome Oncology LLC, Johnson City, New York
  - Winthrop University Hospital, Mineola, New York
  - Clinical Research Alliance, Inc., New Hyde Park, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Texas Oncology - Midland Allison Cancer Center, Midland, Texas
  - US Oncology, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Fairfax Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Roanoke, Virginia
  - MultiCare Regional Cancer Center - Auburn, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Yes
  Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Spigel D, Jotte R, Nemunaitis J, Shum M, Schneider J, Goldschmidt J, Eisenstein J, Berz D, Seneviratne L, Socoteanu M, Bhanderi V, Konduri K, Xia M, Wang H, Hozak RR, Gueorguieva I, Ferry D, Gandhi L, Chao BH, Rybkin I. Randomized Phase 2 Studies of Checkpoint Inhibitors Alone or in Combination With Pegilodecakin in Patients With Metastatic NSCLC (CYPRESS 1 and CYPRESS 2). J Thorac Oncol. 2021 Feb;16(2):327-333. doi: 10.1016/j.jtho.2020.10.001. Epub 2020 Nov 6. PMID 33166722
- [Derived] Albrethsen M, Creeden J, Morand S, DeBiase J, Berry B, Stanbery L, Edelman G, Nemunaitis J. Relationship of hypothyroidism and immune response to pegylated IL-10/nivolumab. Immunotherapy. 2020 Oct;12(14):1041-1046. doi: 10.2217/imt-2020-0016. Epub 2020 Aug 18. PMID 32808556

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completer's included participants who had progression free survival events (Progressive Disease (PD) or death).
Period: Overall Study
Arm/Group | Pegilodecakin+Nivolumab | Nivolumab
Started | 27 | 25
Received at Least 1 Dose of Study Drug | 27 | 24
Completed | 21 | 13
Not Completed | 6 | 12
Not completed — Physician Decision | 0 | 1
Not completed — Sponsor Decision | 6 | 6
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Pegilodecakin + Nivolumab: Participants received Pegilodecakin subcutaneously at 0.8 mg (≤80 kg body weight) or 1.6 mg (>80 kg body weight) once daily in the abdomen, thigh or back of upper arm.
  Nivolumab administered on day 1 of each 14 or 28 day cycle over approximately 30 minutes IV infusion at 240 mg Q2W, or 480 mg Q4W.
- Nivolumab: Participants received Nivolumab on day 1 of each 14 or 28 day cycle over approximately 30 minutes IV infusion at 240 mg Q2W, or 480 mg Q4W.
- Total: Total of all reporting groups
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.2) | 65.9 (10.4) | 67.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 23 | 20 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Objective response rate is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: From Date of Randomization to Progressive Disease, Death from Any cause (Up to 6 months after the last participant randomized)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pegilodecakin + Nivolumab: Participants received Pegilodecakin subcutaneously at 0.8 mg (≤80 kg body weight) or 1.6 mg (>80 kg body weight) once daily in the abdomen, thigh or back of upper arm.
  Nivolumab administered on day 1 of each 14 or 28 day cycle over approximately 30 minutes IV infusion at 240 mg Q2W or 480 mg Q4W.
- Nivolumab: Participants received Nivolumab on day 1 of each 14 or 28 day cycle over approximately 30 minutes IV infusion at 240 mg Q2W or 480 mg Q4W.
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
Number analyzed (Participants) | 27 | 25
Percentage of participants | 14.8 [4.2 to 33.7] | 12.0 [2.6 to 31.2]
Statistical Analysis 1: Comparison: Pegilodecakin + Nivolumab vs Nivolumab; Test type: Superiority; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.3 to 5.9] — Odds Ratio stratified based on tumor histology at randomization (interactive web response system (IWRS)), smoking status (IWRS). Confidence intervals were based on the Clopper-Pearson method

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first day of therapy to the date of death from any cause. Participants who were alive at the end of the follow-up period or were lost to follow-up, OS was censored on the last date the participant was known to be alive.
Time Frame: From Date of Randomization to Death Due to Any Cause (Up to 6 months after the last participant randomized)
Population: All randomized participants. Participants censored: Pegilodecakin + Nivolumab = 6 and Nivolumab = 5.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
Number analyzed (Participants) | 27 | 25
Months | 1.87 [1.51 to 3.58] | 1.94 [1.71 to 2.17]
Statistical Analysis 1: Comparison: Pegilodecakin + Nivolumab vs Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.519 to 1.951] — The estimate of the hazard ration (HR) stratified based on tumor histology at randomization (interactive web response system (IWRS)) and smoking status (IWRS)

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the day of randomization to the first evidence of progression as defined by Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) criteria or death from any cause. Progressive Disease (PD) is a 20% increase over the smallest sum of target lesions or new lesions. Participants who died without a reported prior disease progression were considered to have progressed on the day of their death. Participants who did not progress and were subsequently lost to follow-up had their data censored at the day of last tumor assessment.
Time Frame: From Date of Randomization to Progressive Disease or Death Due to Any Cause (Up to 6 months after the last participant randomized)
Population: All randomized participants. Participants censored: Pegilodecakin + Nivolumab = 12 and Nivolumab = 16.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
Number analyzed (Participants) | 27 | 25
Months | 6.70 [3.09 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate. | 10.74 [4.21 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate.
Statistical Analysis 1: Comparison: Pegilodecakin + Nivolumab vs Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.871, 95% CI 2-sided [0.772 to 4.532]; The estimate of the hazard ration (HR) stratified based on tumor histology at randomization (IWRS) and smoking status (IWRS)

4. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Disease control rate (DCR) is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of Randomization to Objective Progressive Disease or Start of New Anti-Cancer Therapy (Up to 6 Months after the last participant randomization)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
Number analyzed (Participants) | 27 | 25
Percentage of participants | 37.0 [19.4 to 57.6] | 28.0 [12.1 to 49.4]
Statistical Analysis 1: Comparison: Pegilodecakin + Nivolumab vs Nivolumab; Test type: Superiority; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.4 to 4.1] — Odds Ratio stratified based on tumor histology at randomization (IWRS) and smoking status (IWRS). Confidence intervals were based on the Clopper-Pearson method

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST 1.1, or the date of death from any cause in the absence of objectively determined disease progression or recurrence. Participants known to be alive and without disease progression will be censored at the time of the last adequate tumor assessment.
Time Frame: From Date of Randomization to Death Due to Any Cause (Up to 6 months after the last participant randomized)
Population: All randomized participants who received at least one dose of study drug and had CR or PR responses. Participants censored: Pegilodecakin + Nivolumab = 3 and Nivolumab = 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
Number analyzed (Participants) | 4 | 3
Months | NA [7.36 to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate. | 3.06 [1.87 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate.

ADVERSE EVENTS:
Time Frame: Up to 23 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Pegilodecakin + Nivolumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 15/27 | 12/24
Serious Adverse Events (participants affected / at risk) | 13/27 | 9/24
Other Adverse Events (participants affected / at risk) | 27/27 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegilodecakin + Nivolumab (N=27) | Nivolumab (N=24)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Bezoar (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pegilodecakin + Nivolumab (N=27) | Nivolumab (N=24)
Anaemia (Blood and lymphatic system disorders) | 14 (37) | 5 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (15) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (5)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 7 (8) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (7)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Asthenia (General disorders) | 4 (9) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 17 (35) | 10 (18)
Gait disturbance (General disorders) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Injection site rash (General disorders) | 5 (5) | 0 (0)
Oedema peripheral (General disorders) | 4 (11) | 3 (3)
Pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 8 (14) | 4 (4)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (5)
Vaginal infection (Infections and infestations) | 0/10 (0) | 1/11 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (6)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 2 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 4 (5) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 5 (6) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (8) | 3 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (8) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7) | 4 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 7 (10) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1/17 (1) | 0/14 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 10 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 7 (9) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03382912/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03382912/SAP_001.pdf